CLINICAL TRIAL: NCT00624286
Title: A 12-week Treatment, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Assess the Efficacy and Safety of Indacaterol (150 μg o.d.) in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy and Safety of Indacaterol in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2346; EUDRACT Number: 2008-000301-11
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Results first posted 2011-08-18 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; COPD; indacaterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indacaterol 150 μg (Experimental): Patients inhaled indacaterol 150 μg once daily in the morning between 8:00 AM and 11:00 AM via a single-dose dry-powder inhaler (SDDPI) for 12 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol 150 μg
- Placebo to indacaterol (Placebo Comparator): Patients inhaled placebo to indacaterol once daily in the morning between 8:00 AM and 11:00 AM via a single-dose dry-powder inhaler (SDDPI) for 12 weeks. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Placebo to indacaterol

INTERVENTIONS:
Drug: Indacaterol 150 μg — Indacaterol was supplied in powder filled capsules together with a single-dose dry-powder inhaler (SDDPI) device.
  Arms: Indacaterol 150 μg
Drug: Placebo to indacaterol — Placebo to indacaterol was supplied in powder filled capsules together with a single-dose dry-powder inhaler (SDDPI) device.
  Arms: Placebo to indacaterol

SUMMARY:
This study was designed to provide 12 weeks efficacy and safety data of the 150 μg once-daily (od) dose of indacaterol in chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

• Male or female patients aged 40 years or over with moderate to severe chronic obstructive pulmonary disease (COPD) plus

* 20 pack-year smoking history
* Signed informed consent
* Post-bronchodilator forced expiratory volume in 1 second )FEV1) ≥ 30% and < 80% predicted FEV1/FVC (forced vital capacity) < 70%

Exclusion Criteria include:

* History of asthma
* Prior exposure to indacaterol
* Active cancer or history of cancer
* Patients with concomitant pulmonary disease
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Patients with a history of long QT syndrome or whose QTc interval (Bazett's) measured at screening or randomization is prolonged
* Patients unable to successfully use a dry-powder inhaler device or perform spirometry measurements

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (111):
- United States (109):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Jasper, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigator Site, Glendale, Arizona
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Pine Bluff, Arkansas
  - Novartis Investigative Site, Buena Park, California
  - Novartis Investigative Site, Encinitas, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Palmdale, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, San Jose, California
  - Novartis Investigative Site, San Mateo, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Vista, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Fort Collins, Colorado
  - Novartis Investigative Site, Golden, Colorado
  - Novartis Investigator Site, Wheat Ridge, Colorado
  - Novartis Investigative Site, Newark, Delaware
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Largo, Florida
  - Novartis Investigative Site, Ocala, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Rockledge, Florida
  - Novartis Investigator Site, Sarasota, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Zephyrhills, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Austell, Georgia
  - Novartis Investigative Site, Normal, Illinois
  - Novartis Investigative Site, O'Fallon, Illinois
  - Novartis Investigative Site, River Forest, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Ames, Iowa
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, Shawnee, Kansas
  - Novartis Investigative Site, Crescent Springs, Kentucky
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Madisonville, Kentucky
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, Opelousas, Louisiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Clarkston, Michigan
  - Novartis Investigative Site, Flint, Michigan
  - Novartis Investigative Site, Livonia, Michigan
  - Novartis Investigative Site, Troy, Michigan
  - Novartis Investigator Site, Edina, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigator Site, St Louis, Missouri
  - Novartis Investigative Site, Kalispell, Montana
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Cherry Hill, New Jersey
  - Novartis Investigative Site, Summit, New Jersey
  - Novartis Investigative Site, Cortland, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigator Site, Cincinnati, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Thornville, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Erie, Pennsylvania
  - Novartis Investigative Site, Homestead, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Cumberland, Rhode Island
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Gaffney, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, North Charleston, South Carolina
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Union, South Carolina
  - Novartis Investigative Site, Johnson City, Tennessee
  - Novartis Investigative Site, Amarillo, Texas
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, New Braunfels, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Payson, Utah
  - Novartis Investigative Site, Abingdon, Virginia
  - Novartis Investigative Site, Lynchburg, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Spokane Valley, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Morgantown, West Virginia
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Novartis Investigative Site, Lanaken, Belgium
- Novartis Investigator Site, Tauranga, New Zealand

REFERENCES:
- [Derived] Jones PW, Donohue JF, Nedelman J, Pascoe S, Pinault G, Lassen C. Correlating changes in lung function with patient outcomes in chronic obstructive pulmonary disease: a pooled analysis. Respir Res. 2011 Dec 29;12(1):161. doi: 10.1186/1465-9921-12-161. PMID 22206353
- [Derived] Bleecker ER, Siler T, Owen R, Kramer B. Bronchodilator efficacy and safety of indacaterol 150 mug once daily in patients with COPD: an analysis of pooled data. Int J Chron Obstruct Pulmon Dis. 2011;6:431-8. doi: 10.2147/COPD.S21073. Epub 2011 Aug 18. PMID 22003288
- [Derived] Feldman G, Siler T, Prasad N, Jack D, Piggott S, Owen R, Higgins M, Kramer B; INLIGHT 1 study group. Efficacy and safety of indacaterol 150 microg once-daily in COPD: a double-blind, randomised, 12-week study. BMC Pulm Med. 2010 Mar 8;10:11. doi: 10.1186/1471-2466-10-11. PMID 20211002

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol 150 μg | Placebo to Indacaterol
Started | 211 | 205
Completed | 186 | 178
Not Completed | 25 | 27
Not completed — Protocol Deviation | 7 | 9
Not completed — Adverse Event | 6 | 3
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 3 | 2
Not completed — Administrative problems | 3 | 0
Not completed — Lack of Efficacy | 1 | 6
Not completed — Not stated | 0 | 1
Not completed — Abnormal test procedure result(s) | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 150 μg | Placebo to Indacaterol | Total
Number analyzed (Participants) | 211 | 205 | 416
Age Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.89) | 63.2 (9.62) | 63.0 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 95 | 198
  Male | 108 | 110 | 218

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose at the End of the Study (Week 12 + 1 Day, Day 85)
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the average of measurements made 23 hours 10 minutes and 23 hours 45 minutes post-dose at the end of treatment. The analysis included baseline FEV1, FEV1 pre-dose and 30 minutes post-dose of salbutamol during screening, and FEV1 pre-dose and 1 hour post-dose of ipratropium during screening as covariates.
Time Frame: 24 hours post-dose at the end of the study (Week 12 + 1 day, Day 85)
Population: Intent-to-treat population: All randomized patients who received at least 1 dose of study drug, last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg | Placebo to Indacaterol
Number analyzed (Participants) | 201 | 189
Liters | 1.48 (0.018) | 1.35 (0.019)

2. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) 24 Hours Post-dose on Day 2
Description: as for outcome 1
Time Frame: 24 hours post-dose on Day 2
Population: Intent-to-treat population: All randomized patients who received at least 1 dose of study drug. FEV1 data taken within 6 h of rescue medication was excluded from this analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg | Placebo to Indacaterol
Number analyzed (Participants) | 205 | 197
Liters | 1.47 (0.014) | 1.38 (0.014)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Safety population included all patients who received at least one dose of study drug.
Arm/Group | Indacaterol 150 μg | Placebo to Indacaterol
Serious Adverse Events (participants affected / at risk) | 7/211 | 5/205
Other Adverse Events (participants affected / at risk) | 30/211 | 37/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=211) | Placebo to Indacaterol (N=205)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haematoma (Vascular disorders) | 1 | 0
Vascular pseudoaneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=211) | Placebo to Indacaterol (N=205)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 18 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.